CLINICAL TRIAL: NCT03752996
Title: ACURATE TF™ Transfemoral Aortic Bioprosthesis for Implantation in Patients With Severe Aortic Stenosis
Brief Title: ACURATE TF™ Transfemoral Aortic Bioprosthesis for Implantation in Patients With Severe Aortic Stenosis (2011-03)
Acronym: 2011-03
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Symetis SA (Industry)
Responsible Party: Sponsor
Organization: Boston Scientific Corporation (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-03
Record Dates: First submitted 2018-11-21; First posted 2018-11-26 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Aortic Stenosis Symptomatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ACURATE TF™ Aortic Valve System (Experimental): ACURATE TF™ Aortic Valve System is intended for subjects with severe symptomatic Aortic Stenosis and considered high risk for surgical conventional Aortic Valve Replacement .
  Interventions: Device: ACURATE TF™ Aortic Valve System

INTERVENTIONS:
Device: ACURATE TF™ Aortic Valve System — Transcatheter Aortic Valve Implantation

SUMMARY:
First-In-Man Study on the ACURATE TF™ Transfemoral Aortic Bioprosthesis Implantation in Patients with Severe Aortic Stenosis to collect human feasibility data pertaining to the safety and performance of the device.

DETAILED DESCRIPTION:
A single arm, prospective, multicenter, non-randomized, open trial, up to 5 Years follow-up with the Symetis ACURATE TF™ Transfemoral Aortic Bioprosthesis for minimal invasive implantation via transfemoral access to treat patients with severe aortic stenosis where conventional aortic valve replacement (AVR) via open heart surgery is considered to be associated with high risk.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 75 years of age and older
2. Logistic EuroSCORE ≥ 20%
3. Severe aortic stenosis characterized by mean aortic gradient > 40 mmHg or peak jet velocity > 4.0 m/s or aortic valve area < 1.0 cm2
4. New York Heart Association (NYHA) Functional Class > II
5. Aortic annulus diameter from ≥ 21mm up to ≤ 27mm measured by TEE
6. Patient not a surgical candidate due to significant co-morbid conditions unrelated to aortic stenosis
7. Patient willing to participate in the study and provide signed informed consent

Exclusion Criteria:

1. Unicuspid or bicuspid aortic valve
2. Extreme eccentricity of calcification
3. Severe mitral regurgitation ( >2+)
4. Pre-existing prosthetic heart valve in any position and / or prosthetic ring
5. Aortic or peripheral anatomy NOT appropriate for transfemoral implant
6. Thoracic (TAA) or abdominal (AAA) aortic aneurysm
7. Presence of endovascular stent graft for treatment of TAA or AAA
8. Trans-esophageal echocardiogram (TEE) is contraindicated
9. Left Ventricle Ejection Fraction (LVEF) < 30% by echocardiography (ECHO)
10. ECHO evidence of intracardiac mass, thrombus, or vegetation
11. Acute Myocardial Infarction (AMI) within 1 month prior to implant procedure
12. Percutaneous Coronary Intervention (PCI), except for balloon valvuloplasty (BAV) within 1 month prior to implant procedure
13. Previous Transient Ischemic Attack (TIA) or stroke within 3 months prior to implant procedure
14. Active ulcer or gastrointestinal (GI) bleeding within 3 months prior to implant procedure
15. Any scheduled surgical or percutaneous procedure to be performed prior to 30 day visit
16. History of bleeding diathesis or coagulopathy or refusal of blood transfusions
17. Systolic pressure <80 mmHg, cardiogenic shock, need for inotropic support or Intra-Aortic Balloon Pump (IABP)
18. Primary hypertrophic obstructive cardiomyopathy (HOCM)
19. Active infection, endocarditis or pyrexia
20. Hepatic failure
21. Chronic renal dysfunction with serum creatinine > 2.5 mg/dL or renal dialysis
22. Refusal of surgery
23. Severe Chronic Obstruction Pulmonary Disease (COPD) requiring home oxygen
24. Neurological disease severely affecting ambulation or daily functioning, or dementia
25. Life expectancy < 12 months due to non-cardiac co-morbid conditions
26. Known hypersensitivity/contraindication to study medication, contrast media, or nitinol
27. Currently participating in an investigational drug or another device study

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 140 (Actual)
Dates: Start 2012-05-09 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Freedom from all-cause mortality | 30-Days
  Rate of all-cause mortality

SECONDARY OUTCOMES:
Rate of MACCE (major cardiac and cerebrovascular event) | 30-Days and 12-Months
  Rate of major cardiac and cerebrovascular event (MACCE) defined as cardiovascular death, myocardial infarction and stroke

CONTACTS AND LOCATIONS:
Overall Officials: Won Keun Kim, Dr. Med., Principal Investigator — Kerckhoff Klinik Bad Nauheim, Germany
Locations (5):
- Instituto Dante Pazzanese de Cardiologia, São Paulo, Brazil
- Germany (4):
  - Kerckhoff Klinik GmbH, Bad Nauheim
  - Universitätsklinikum Bonn, Bonn
  - Herzzentrum Universitätsklinikum Köln, Cologne
  - Universitäres Herzzentrum Hamburg, Hamburg

IPD SHARING:
Plan to Share IPD: No